CLINICAL TRIAL: NCT04131049
Title: Comparison of Carbohydrate Counting and Food Insulin Index Methods in the Determination of Insulin Doses for High- and Low-Glycemic Index Meals in Adolescents With Type 1 Diabetes
Brief Title: Comparison of Two Different Insulin Dose Calculation Algorithms in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zeynep Caferoglu, PhD, Assistant Professor Doctor, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 8811
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Insulin-Dependent Diabetes Mellitus 1
Keywords: Adolescent; Carbohydrate Counting; Food Insulin Index; Glycemic Index; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate Counting (Experimental): The insulin doses of the breakfasts were calculated according to carbohydrate counting.
  Interventions: Other: High GI calculated by CC (CHGI); Other: Low GI calculated by CC (CLGI)
- Food Insulin Index (Experimental): The insulin doses of the breakfasts were calculated according to food insulin index.
  Interventions: Other: High GI calculated by FII (FHGI); Other: Low GI calculated by FII (FLGI)

INTERVENTIONS:
Other: High GI calculated by CC (CHGI) — This test meal with high GI were served as a breakfast after 8-hours fasting and participants were asked to consume the meal in full, within 20 min.
  Arms: Carbohydrate Counting
Other: Low GI calculated by CC (CLGI) — This test meal with low GI were served as a breakfast after 8-hours fasting and participants were asked to consume the meal in full, within 20 min.
  Arms: Carbohydrate Counting
Other: High GI calculated by FII (FHGI) — This test meal with high GI were served as a breakfast after 8-hours fasting and participants were asked to consume the meal in full, within 20 min.
  Arms: Food Insulin Index
Other: Low GI calculated by FII (FLGI) — This test meal with low GI were served as a breakfast after 8-hours fasting and participants were asked to consume the meal in full, within 20 min.
  Arms: Food Insulin Index

SUMMARY:
The aim of this study is to compare the impact of carbohydrate counting (CC) method which is standard insulin dose calculation algorithm and food insulin index (FII) method which is a new algorithm on postprandial glucose following a high fat and a high protein meal in adolescent with type 1 diabetes. A randomized, single-blind and crossover trial included 14 adolescents aged 14-18 years with type 1 diabetes. All participants were sent to their homes for 4 consecutive days with a different glycemic index breakfast. The insulin doses of the meals were calculated according to CC and FII methods. Test breakfasts with different GIs and insulin requirements calculated with different algorithms are as follows: High GI calculated by CC (CHGI), low GI calculated by CC (CLGI), high GI calculated by FII (FHGI) and low GI calculated by FII (FLGI).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 14-18 years adolescents
* Type 1 diabetes diagnosed for at least one year
* Performing self-monitoring of blood glucose and doses of insulin at least four times daily
* HbA1c ≤ 9.6% for the last three months
* Negative fasting C-peptide (<0.1 nmol/L)
* Total daily insulin use of ≥ 0.5 U/kg
* World Health Organization BMI/age z-score of -1 to below 3

Exclusion Criteria:

* Complications of diabetes or other medical conditions including celiac disease
* Treatment with oral hypoglycaemic agents
* Food allergies, intolerances, or eating disorder
* Intestinal malabsorptions
* Delayed gastric emptying
* Viral or bacterial infection
* Physical or mental disability
* Clinical condition related to impaired digestive system such as cystic fibrosis

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose response by glucometer | Four hours postprandial period (from fasting to 240 minutes after the test breakfast)
  Postprandial glucose response was quantified as incremental area under the curve (iAUC) (mg/dL x minutes), which was calculated according to the trapezoidal rule by using blood glucose values at time points 0, 30, 60, 90, 120, 150, 180, 210 and 240 minutes.
Postprandial glucose response by continous glucose monitoring | Four hours postprandial period (from fasting to 240 minutes after the test breakfast)
  Postprandial glucose response was quantified as incremental area under the curve (iAUC) (mg/dL x minutes), which was calculated according to the trapezoidal rule by using blood glucose values at time points 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 65, 70, 75, 80, 85, 90, 95, 100, 105, 110, 115, 120, 125, 130, 135, 140, 145, 150, 155, 160, 165, 170, 175, 180, 185, 190, 195, 200, 205, 210, 215, 220, 225, 230, 235 and 240 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Health Sciences, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Erdal B, Caferoglu Z, Hatipoglu N. The comparison of two mealtime insulin dosing algorithms for high and low glycaemic index meals in adolescents with type 1 diabetes. Diabet Med. 2021 Mar;38(3):e14444. doi: 10.1111/dme.14444. Epub 2020 Dec 20. PMID 33119135

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT04131049/Prot_SAP_000.pdf